CLINICAL TRIAL: NCT04103671
Title: Micro-invasive Pars-plana Vitrectomy vs Panretinal Photocoagulation for Severe Non-Proliferative Diabetic Retinopathy A Randomized Clinical Trial
Brief Title: Pars-plana Vitrectomy vs Panretinal Photocoagulation for Severe NPDR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019KYPJ108
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Non Proliferative Diabetic Retinopathy
Keywords: NPDR; Pars-plana vitrectomy; panretinal photocoagulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Prompt panretinal photocoagulation
  Interventions: Procedure: Prompt panretinal photocoagulation
- Group B (Experimental): Micro-invasive Pars-plana vitrectomy
  Interventions: Procedure: 25G Pars-plana vitrectomy

INTERVENTIONS:
Procedure: Prompt panretinal photocoagulation — Study eyes that receive panretinal photocoagulation (prompt PRP eyes at baseline) should have 1200 to1600 burns with a spot size on the retina of approximately 500 microns given over 1 to 3 sittings and completed within 4 weeks of initiation
  Arms: Group A
Procedure: 25G Pars-plana vitrectomy — Study eyes that receive standard 25G Pars-plana vitrectomy that remove all the vitreous, without laser or Silicone oil tamponade, but filled with perfusion fluid. Surgery should be completed within 4 weeks after randomization.
  Arms: Group B

SUMMARY:
It is estimated that there are about 600 million diabetes mellitus (DM) patients all over the world until 2040，and almost 50% of whom have some degree of diabetic retinopathy (DR) at any given time. About 5% to 10% diabetic retinopathy would develop vision-threatening complications, including proliferative diabetic retinopathy (PDR), capillary non-perfusion, or macular edema. Data from the DRS suggest that given long enough duration of diabetes, approximately 60% of patients with DR will develop PDR, and without intervention, 75% nonproliferative diabetic retinopathy (NPDR) will development PDR within 1 year follow up, 45% will develop high-risk PDR, nearly half of PDR will experience profound visual loss. panretinal photocoagulation (PRP) only reduced 50% risk of sever visual loss and about 25% of the sNPDR patients who finished PRP need Pars-plana vitrectomy (PPV) in a 5 year follow up.

Vitreous have been proven to play an important role in the development of NPDR to PDR, which were the collection of vascular endothelial growth factor (VEGF) factors and the major component of proliferative lesion in the later stage of PDR.

Micro-invasive Pars-plana vitrectomy has been shown as a safe and effective method in the treatment of PDR, through removing the pathological vitreous, proliferative membrane and also the VEGF factors. However, whether or not Micro-invasive Pars-plana vitrectomy will be more effective than PRP to control the progression of NDPR remained unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years, male or female
2. Type 1 or type 2 diabetes
3. Presence of severe NPDR according to the diagnosis of 4-2-1 rule,

   One or more of the following, in the absence of PDR:
   * More than 20 intraretinal hemorrhages in each of four quadrants
   * Definite venous beading in two or more quadrants
   * Prominent intraretinal microvascular abnormality (IRMA) in one or more quadrants
4. Best corrected Electronic-Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity letter score > 24 (approximate Snellen equivalent 20/320) on the day of randomization.
5. Media clarity, pupillary dilation, and study participant cooperation sufficient to administer PRP and obtain adequate fundus photographs and optical coherence tomography (OCT).
6. Able and willing to provide informed consent

Exclusion Criteria:

1. Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant
2. In the opinion of the investigator, A condition that would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
3. Participation in an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval for the indication being studied.
4. Blood pressure > 180/110 (systolic above 180 or diastolic above 110).

   *If blood pressure is brought below 180/110 by anti-hypertensive treatment, individual can become eligible.
5. Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization
6. Systemic anti-VEGF or pro-VEGF treatment within 4 months prior to randomization

   * These drugs should not be used during the study
7. For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 3 years.

   * Women who are potential study participants should be questioned about the potential for pregnancy. Investigator judgment is used to determine when a pregnancy test is needed
8. History of prior panretinal photocoagulation (prior PRP is defined as ≥100 burns outside of the posterior pole
9. If macular edema is present, it is considered to be primarily due to a cause other than diabetic macular edema.
10. An ocular condition is present (other than diabetic retinopathy) that, in the opinion of the investigator, might alter visual acuity during the course of the study (e.g., retinal vein or artery occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.).
11. Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye were otherwise normal).
12. History of intravitreal anti-VEGF treatment at any time in the past 2 months
13. History of corticosteroid treatment (intravitreal or peribulbar) at any time in the past 4 months.
14. History of major ocular surgery (including vitrectomy, cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months or anticipated within the next 6 months following randomization.
15. History of laser capsulotomy performed within 2 months prior to randomization
16. Aphakia.
17. Uncontrolled glaucoma (in investigator's judgment).
18. Exam evidence of severe external ocular infection, including conjunctivitis, chalazion, or substantial blepharitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
progression rate of severe non proliferative diabetic retinopathy | 12 months
  the number of patients with severe non proliferative diabetic retinopathy progressed to proliferative diabetic retinopathy in each group from the baseline to 12 months

SECONDARY OUTCOMES:
the change of best corrected visual acuity | 12 months
  The mean change in best corrected visual acuity in each group from baseline to 12 months
the rate of re-treatment | 12 months
  The number of patients who need re-treatment including supplement laser or vitrectomy from baseline to 12 months
The occurrence of diabetic macular edema | 12 months
  The occurrence number of diabetic macular edema in each group from baseline to 12 months
The change of central retinal thickness | 12 months
  the change of central retinal thickness from baseline to 12 months
The change of visual field | 12 months
  the change of visual field from baseline to 12 months
The occurrence of cataract | 12 months
  the occurrence of cataract from baseline to 12 months
The change of quality of life | 12 months
  the change of quality of life as assessed by questionnaire at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng W, Chen S, Ding X, Lai K, Xiao S, Lin Y, Liu B, Jin L, Li J, Wu Y, Ma Y, Lu L, Liu Y, Li T. Microinvasive pars plana vitrectomy versus panretinal photocoagulation in the treatment of severe non-proliferative diabetic retinopathy (the VIP study): study protocol for a randomised controlled trial. BMJ Open. 2021 Feb 22;11(2):e043371. doi: 10.1136/bmjopen-2020-043371. PMID 33619191